CLINICAL TRIAL: NCT06520319
Title: Head-to-head Study of 68Ga-MGS5 Versus 68Ga-DOTATATE PET/CT in Patients With Medullary Thyroid Carcinoma: a Prospective Study
Brief Title: Head-to-head Study of 68Ga-MGS5 Versus 68Ga-DOTATATE PET/CT in Patients With Medullary Thyroid Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, Director, Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian-68Ga-MGS5
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Medullary Thyroid Carcinoma
MeSH Terms: conditions — Carcinoma, Medullary | interventions — gallium Ga 68 dotatate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients will undergo a 68Ga-MGS5 PET/CTF and 68Ga-DOTATATE PET/CT (Experimental): MTC Patients received 68Ga-DOTATATE PET/CT imaging and a single injection of 68Ga-MGS5 and two PET/CT scans 1 hour and 2 hours after the injection within one week.
  Interventions: Drug: 68Ga-MGS5

INTERVENTIONS:
Drug: 68Ga-MGS5 — Each patient received a single intravenous injection of 68Ga-DOTATATE (2-4 mCi) and underwent PET/CT scanning 40-60 minutes after the injection. Or receive one intravenous injection of 68Ga-MGS5 and undergo two PET/CT scans at 1 and 2 hours post-injection, respectively.
  Other Names: 68Ga-DOTATATE

SUMMARY:
Cholecystokinin-2 (CCK2) receptor is overexpressed in more than 90% of MTC cases, and preclinical studies have shown that 68Ga-MGS5 (targeting CCK2) has good stability in vivo and is promising for diagnosis and staging of MTC. This prospective study will compare the diagnostic effects of 68Ga-MGS5 and 68Ga-DOTATATE on MTC primary foci, lymph node metastasis, and distant metastasis, and explore the effect of 68Ga-MGS5 PET/CT on the clinical staging (TNM staging) of MTC.

DETAILED DESCRIPTION:
This study was planned to enroll 20 patients with suspected MTC and MTC recurrence who attended the First Hospital of Fujian Medical University from June 2023 onwards. Each patient completed PET/CT examination within 1 week, one 68Ga-DOTATATE PET/CT whole-body examination and two 68Ga-MGS5 PET/CT whole-body examinations (1 hour and 2 hours after injection, respectively). CCK2 immunohistochemical staining and expression scoring of primary foci and lymph node metastases were also performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender, aged ≥ 18 years and ≤80 years.
* Patients with pathologic findings confirming the diagnosis of MTC
* Patients with MTC recurrence
* Signed written consent

Exclusion Criteria:

* Pregnant or breastfeeding female patients
* Patients with claustrophobic behavior
* The inability or unwillingness of the research participant, parent or legal representative to provide written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
SUVmax and SUVpeak | through study completion, an average of 2 years
  Determination of SUVmean and SUVpeak for detected lesions and discernible organs of 68Ga-MGS5 and 68Ga-DOTATATE scan.

SECONDARY OUTCOMES:
immunohistochemistry | through study completion, an average of 2 years
  Primary and lymph node metastases were stained with CCK2 immunohistochemistry and scored.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No